CLINICAL TRIAL: NCT02996643
Title: Determine the Optimum Applied Pressure for the Brace Treatment of Scoliosis
Brief Title: Ultrasound-Assisted Brace Casting for AIS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro000028133
Record Dates: First submitted 2016-12-09; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Scoliosis; Adolescence
Keywords: Adolescent Idiopathic Scoliosis; Brace Treatment; Ultrasound Imaging
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional method (No Intervention): The traditional brace design method will be used to design a spinal brace.
- Intervention (Active Comparator): A custom Providence brace standing frame, a medical ultrasound system, a custom pressure measurement system, and in-house Ultrasound measurement software were used to assist brace casting for the intervention group.
  Interventions: Device: Ultrasound Assisted Group

INTERVENTIONS:
Device: Ultrasound Assisted Group — A custom brace standing frame, a medical ultrasound system, a custom pressure measurement system, and in-house Ultrasound measurement software were used to assist brace casting for the intervention group.
  Arms: Intervention

SUMMARY:
Adolescent Idiopathic Scoliosis (AIS) is a three-dimensional deformity of the spine associated with vertebral rotation. Brace treatment is the most commonly used non-surgical treatment. To obtain the best possible outcome, the best in-brace correction within the patient's accepted tolerance must be provided. However, in the existing clinical practice, the immediate in-brace correction cannot be measured during the design and fitting of the brace because the correction is determined using a radiograph. This study is to evaluate the effect of applying ultrasound to measure the stimulated in-brace correction during brace casting.

DETAILED DESCRIPTION:
Background: Adolescent Idiopathic Scoliosis (AIS) is a three-dimensional deformity of the spine associated with vertebral rotation. Brace treatment is the most commonly used non-surgical treatment. To obtain the best possible outcome, the best in-brace correction within the patient's accepted tolerance must be provided. However, in the existing clinical practice, the immediate in-brace correction cannot be measured during the design and fitting of the brace because the correction is determined using a radiograph.

Objectives: The objective of this study is to use ultrasound method to determine the optimum tolerable applied pressure level that can provide maximum in-brace correction.

Procedure:

Control Group: In the traditional method, each brace will be constructed using a plaster cast of the patient's trunk. Before the plaster cast hardens, the subject will lie on a casting board with multiple brace pads applied to correct the curve(s). The trim lines, pad placement, and areas of relief are then determined by the orthotist and guided by the curvature seen on the pre-brace PA spine radiograph.

Intervention Group: Before applying the plaster, subjects will lie on the custom designed frame. Two ultrasound scans will be performed and the average Cobb value will be used as the baseline. Multiple adjustable brace pads, each allowing for 6° of freedom and variable forces, will be applied to the patients' body according to orthotist suggestion. The apical brace pad that is used to control the major curve will be marked relative to the casting board as the reference location. The major pressure pad will be moved up 1 inch, then down 1 inch relative to the reference location. The 1 inch increment corresponds to the casting board, but finer adjustment is available. Two repeated ultrasound scans will be performed at each pad location (total 3 locations), and the average in-brace Cobb values will be estimated to determine optimum apical brace pad location. Next, pressure will be increased incrementally up to the tolerance level of the subject; this will be done by inflating the bladder at the apical brace pad. Another two ultrasound scans will then be performed to confirm that the maximum in-brace Cobb value is obtained. The orthotist will use this configuration to set the pad size and location once the plaster cast has been applied.

ELIGIBILITY:
Inclusion Criteria:

* AIS patients who are prescribed braces to treat their spinal deformity.

Exclusion Criteria:

* Any one does not want to participate.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2012-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
In-brace Cobb angle | 6 weeks
  In-brace radiographs will be obtained after patients use their braces for 6 weeks

SECONDARY OUTCOMES:
Number of adjustments | 6 weeks
  Check if brace adjustment is required

CONTACTS AND LOCATIONS:
Overall Officials: Edmond Lou, PhD, Principal Investigator — University of Alberta
Locations (1):
- Medicine and Dentistry, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lou EH, Hill DL, Donauer A, Tilburn M, Hedden D, Moreau M. Results of ultrasound-assisted brace casting for adolescent idiopathic scoliosis. Scoliosis Spinal Disord. 2017 Aug 8;12:23. doi: 10.1186/s13013-017-0130-2. eCollection 2017. PMID 28795156